CLINICAL TRIAL: NCT05855460
Title: Estimation of the Tissue and Serum Levels of Interleukin (IL) -35 in Mycosis Fungoides: a Case Control Study.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Maha Fathy Elmasry, Maha Fathy Elmasry, MD, Cairo University
Other Study IDs: Yasmfil35
Record Dates: First submitted 2023-05-03; First posted 2023-05-11 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Mycosis Fungoides
MeSH Terms: conditions — Mycosis Fungoides | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Mycosis fungoides patients: Blood sample and skin biopsy for assessment of IL35 by ELISA
  Interventions: Diagnostic Test: Skin biopsy
- Normal healthy controls: Blood sample and skin biopsy for assessment of IL35 levels by ELISA
  Interventions: Diagnostic Test: Skin biopsy

INTERVENTIONS:
Diagnostic Test: Skin biopsy — biochemical assessment for measurement IL35 by ELISA (Enzyme linked immunosorbent assay) technique in tissue and serum samples of all thirty patients and healthy controls.
  Other Names: Blood sample

SUMMARY:
Tissue and serum samples from 20 MF patients and 20 normal healthy controls will be subjected for biochemical assessments by ELISA (Enzyme- linked immune-sorbent assay) for assessing the level of IL35.

DETAILED DESCRIPTION:
Tissue and serum samples from 20 MF patients and 20 normal healthy controls will be subjected for biochemical assessments by ELISA (Enzyme- linked immune-sorbent assay) for assessing the level of IL35

ELIGIBILITY:
Inclusion Criteria:

* Patients with mycosis fungoides. Both genders. Age group ≥ 18 years old.

Exclusion Criteria:

* Patients with any other skin diseases. Patients who received treatments for mycosis fungoides in the past three months.

Subjects with history of solid or hematological malignancy as leukemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with mycosis fungoides. Subjects attending plastic surgery units for abdominoplasty will be enrolled as controls.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-01-12 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
To assess and compare tissue and serum levels of interleukin 35 (IL -35) in mycosis fungoides patients and normal controls. | 1 year
  To assess and compare tissue and serum levels of interleukin 35 (IL -35) in mycosis fungoides patients and normal controls.

SECONDARY OUTCOMES:
Correlating tissue and serum levels of IL-35 in mycosis fungoides patients with patients age, sex, duration, extent and stage of the disease. L | 1 year
  Correlating tissue and serum levels of IL-35 in mycosis fungoides patients with patients age, sex, duration, extent and stage of the disease.

CONTACTS AND LOCATIONS:
Overall Officials: Maha Fathy Elmasry, MD, Principal Investigator — Cairo University
Locations (1):
- Cairo University, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Undecided